CLINICAL TRIAL: NCT06655805
Title: Registry for Automated Mechanical VEntilation in Adults
Acronym: RAVE
Status: Recruiting | Type: Observational
Sponsor: Hamilton Medical AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HM - RAVE
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Insufficiency Requiring Mechanical Ventilation
Keywords: Real world data; Acute respiratory failure; Respiratory support; Invasive Mechanical Ventilation (IMV); Non Invasive Ventilation (NIV); High Flow Nasal Oxygen (HFNO)
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- One cohort of consecutive patients: One cohort of consecutive patients admitted to the intensive care unit while on IMV or in need of HFNO, NIV lung support due to acute respiratory failure.
  Interventions: Device: Non-invasive ventilation, Invasive mechanical ventilation, high-flow nasal oxygen

INTERVENTIONS:
Device: Non-invasive ventilation, Invasive mechanical ventilation, high-flow nasal oxygen — No intervention is intended by the nature of this observational study.

SUMMARY:
The aim of the here proposed study is to assess safety, performance and provide real world evidence (RWE) of the Hamilton Medical AG automated mechanical ventilation software packages in consecutive critically ill patients admitted to the intensive care unit.

DETAILED DESCRIPTION:
The harmful effect of invasive mechanical ventilation can be prevented by intensive training of ICU physicians, respiratory therapists, and ICU nurses on the one hand, and by improvement of the technology installed in ventilators on the other hand. Advanced mechanical ventilation modes use new technologies to assist physiology, optimize gas exchange and minimize ventilator induced lung injury. Modes such as proportional assist ventilation and neuronally adjusted ventilatory assist deliver assisted ventilation proportional to the patient's effort, improving ventilator patient synchrony. The Adaptive Support Ventilation (ASV) mode automatically adjust tidal volume and respiratory rate based on patient's respiratory mechanics to protect from mechanical ventilator induced lung injury, hence deliver safe mechanical ventilation. The implementation of advanced closed-loop systems automates medical reasoning and has potential to improve patient ventilator interactions, the time spent on mechanical ventilation, staff workload and potentially outcome.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years. Any patient in need of HFNO, NIV and IMV at some time during its ICU stay.

Exclusion Criteria:

Expected to be weaned from HFNO, NIV within 2 hours. Expected to be weaned and extubated from IMV without subsequent need of HFNO or NIV support within 2 hours.

Expected to be transferred to another non-participating ICU within 2 hours. Moribund subject: death expected within 2 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to the intensive care unit while on IMV or in need of HFNO, NIV lung support due to acute respiratory failure, or protection of the airway due to a non-respiratory life-threatening condition.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint is determinate by the percentage of breaths outside of the optimal and the acceptable zone during the observation period, based on the following ventilation parameters if available: | Day 0 - Day 7
  Tidal volume (VT), maximum pressure (Pmax), oxygen saturation measured by pulse oximetry (SpO2), end-tidal partial pressure of carbon dioxide (PetCO2), Respiratory rate (RR) for spontaneous breathing subjects, Pmax-PEEP for passive ARDS subjects, driving pressure, mechanical power. The optimal and sub-optimal ranges are defined by current recommendations for different clinical conditions including normal lungs, brain injury, ARDS, and chronic hypercapnia.
The efficiency endpoint is determinate by the percentage of breath inside of the optimal zone during the observation period based on the following ventilation parameters if available: | Day 0 - Day 7
  tidal volume (VT), maximum pressure (Pmax), oxygen saturation measured by pulse oximetry (SpO2), end-tidal partial pressure of carbon dioxide (PetCO2), Respiratory rate (RR) for spontaneous breathing subjects, Pmax-PEEP for passive ARDS subjects, driving pressure, mechanical power. The optimal and sub-optimal ranges are defined by current recommendations for different clinical conditions including normal lungs, brain injury, ARDS, and chronic hypercapnia.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Porta, MD, Principal Investigator — Kantonsspital Chur, Chur, Switerzland 7000
Locations (4):
- Switzerland (4):
  - HOCH Health Ostschweiz, Clinics for Intensive Care Medicine, Surgical ICU, Sankt Gallen, Canton of St. Gallen
  - Kantonsspital Chur, Chur, Kanton Graubünden
  - HOCH Health Ostschweiz, Clinics for Intensive Care Medicine, Medical ICU, Sankt Gallen, St.Gallen
  - Kantonsspital Winterthur, Zentrum für Intensivmedizin, Winterthur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Neto AS, Simonis FD, Barbas CS, Biehl M, Determann RM, Elmer J, Friedman G, Gajic O, Goldstein JN, Linko R, Pinheiro de Oliveira R, Sundar S, Talmor D, Wolthuis EK, Gama de Abreu M, Pelosi P, Schultz MJ; PROtective Ventilation Network Investigators. Lung-Protective Ventilation With Low Tidal Volumes and the Occurrence of Pulmonary Complications in Patients Without Acute Respiratory Distress Syndrome: A Systematic Review and Individual Patient Data Analysis. Crit Care Med. 2015 Oct;43(10):2155-63. doi: 10.1097/CCM.0000000000001189. PMID 26181219
- [Background] Guo L, Wang W, Zhao N, Guo L, Chi C, Hou W, Wu A, Tong H, Wang Y, Wang C, Li E. Mechanical ventilation strategies for intensive care unit patients without acute lung injury or acute respiratory distress syndrome: a systematic review and network meta-analysis. Crit Care. 2016 Jul 22;20(1):226. doi: 10.1186/s13054-016-1396-0. PMID 27448995
- [Background] Campbell RS, Branson RD, Johannigman JA. Adaptive support ventilation. Respir Care Clin N Am. 2001 Sep;7(3):425-40, ix. doi: 10.1016/s1078-5337(05)70049-6. PMID 11517032
- [Background] Linton DM, Potgieter PD, Davis S, Fourie AT, Brunner JX, Laubscher TP. Automatic weaning from mechanical ventilation using an adaptive lung ventilation controller. Chest. 1994 Dec;106(6):1843-50. doi: 10.1378/chest.106.6.1843. PMID 7988211
- [Background] Brunner JX, Iotti GA. Adaptive Support Ventilation (ASV). Minerva Anestesiol. 2002 May;68(5):365-8. PMID 12029247
- [Background] Arnal JM, Wysocki M, Novotni D, Demory D, Lopez R, Donati S, Granier I, Corno G, Durand-Gasselin J. Safety and efficacy of a fully closed-loop control ventilation (IntelliVent-ASV(R)) in sedated ICU patients with acute respiratory failure: a prospective randomized crossover study. Intensive Care Med. 2012 May;38(5):781-7. doi: 10.1007/s00134-012-2548-6. Epub 2012 Mar 30. PMID 22460854
- [Background] Lellouche F, Bouchard PA, Simard S, L'Her E, Wysocki M. Evaluation of fully automated ventilation: a randomized controlled study in post-cardiac surgery patients. Intensive Care Med. 2013 Mar;39(3):463-71. doi: 10.1007/s00134-012-2799-2. Epub 2013 Jan 22. PMID 23338569
- [Background] Babic SA, Chatburn RL. Laboratory Evaluation of Cuff Pressure Control Methods. Respir Care. 2020 Jan;65(1):62-67. doi: 10.4187/respcare.06728. Epub 2019 Jul 30. PMID 31363001
- [Background] Blakeman T, Rodriquez D Jr, Woods J, Cox D, Elterman J, Branson R. Automated control of endotracheal tube cuff pressure during simulated flight. J Trauma Acute Care Surg. 2016 Nov;81(5 Suppl 2 Proceedings of the 2015 Military Health System Research Symposium):S116-S120. doi: 10.1097/TA.0000000000001234. PMID 27602899
- [Background] OTIS AB, FENN WO, RAHN H. Mechanics of breathing in man. J Appl Physiol. 1950 May;2(11):592-607. doi: 10.1152/jappl.1950.2.11.592. No abstract available. PMID 15436363
- [Background] MEAD J. The control of respiratory frequency. Ann N Y Acad Sci. 1963 Jun 24;109:724-9. doi: 10.1111/j.1749-6632.1963.tb13500.x. No abstract available. PMID 13934289
- [Background] Botta M, Wenstedt EFE, Tsonas AM, Buiteman-Kruizinga LA, van Meenen DMP, Korsten HHM, Horn J, Paulus F, Bindels AGJH, Schultz MJ, De Bie AJR. Effectiveness, safety and efficacy of INTELLiVENT-adaptive support ventilation, a closed-loop ventilation mode for use in ICU patients - a systematic review. Expert Rev Respir Med. 2021 Nov;15(11):1403-1413. doi: 10.1080/17476348.2021.1933450. Epub 2021 Jul 31. PMID 34047244
- [Background] Buiteman-Kruizinga LA, Mkadmi HE, Serpa Neto A, Kruizinga MD, Botta M, Schultz MJ, Paulus F, van der Heiden PLJ. Effect of INTELLiVENT-ASV versus Conventional Ventilation on Ventilation Intensity in Patients with COVID-19 ARDS-An Observational Study. J Clin Med. 2021 Nov 19;10(22):5409. doi: 10.3390/jcm10225409. PMID 34830691
- [Background] Chelly J, Mazerand S, Jochmans S, Weyer CM, Pourcine F, Ellrodt O, Thieulot-Rolin N, Serbource-Goguel J, Sy O, Vong LVP, Monchi M. Automated vs. conventional ventilation in the ICU: a randomized controlled crossover trial comparing blood oxygen saturation during daily nursing procedures (I-NURSING). Crit Care. 2020 Jul 22;24(1):453. doi: 10.1186/s13054-020-03155-3. PMID 32698860
- [Background] Arnal JM, Garnero A, Novotni D, Corno G, Donati SY, Demory D, Quintana G, Ducros L, Laubscher T, Durand-Gasselin J. Closed loop ventilation mode in Intensive Care Unit: a randomized controlled clinical trial comparing the numbers of manual ventilator setting changes. Minerva Anestesiol. 2018 Jan;84(1):58-67. doi: 10.23736/S0375-9393.17.11963-2. Epub 2017 Jul 5. PMID 28679200
- [Background] Roca O, Caritg O, Santafe M, Ramos FJ, Pacheco A, Garcia-de-Acilu M, Ferrer R, Schultz MJ, Ricard JD. Closed-loop oxygen control improves oxygen therapy in acute hypoxemic respiratory failure patients under high flow nasal oxygen: a randomized cross-over study (the HILOOP study). Crit Care. 2022 Apr 14;26(1):108. doi: 10.1186/s13054-022-03970-w. PMID 35422002
- [Background] Davidson AC, Banham S, Elliott M, Kennedy D, Gelder C, Glossop A, Church AC, Creagh-Brown B, Dodd JW, Felton T, Foex B, Mansfield L, McDonnell L, Parker R, Patterson CM, Sovani M, Thomas L; BTS Standards of Care Committee Member, British Thoracic Society/Intensive Care Society Acute Hypercapnic Respiratory Failure Guideline Development Group, On behalf of the British Thoracic Society Standards of Care Committee. BTS/ICS guideline for the ventilatory management of acute hypercapnic respiratory failure in adults. Thorax. 2016 Apr;71 Suppl 2:ii1-35. doi: 10.1136/thoraxjnl-2015-208209. No abstract available. PMID 26976648